CLINICAL TRIAL: NCT04241289
Title: Detection and Neurological Impact of Cerebrovascular Events in Cardiac Surgery Patients: A Cohort Evaluation Pilot (NeuroVISION Cardiac Pilot)
Brief Title: Detection and Neurological Impact of Cerebrovascular Events in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroVISION Cardiac Pilot
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Silent Stroke; Cognitive Decline
Keywords: covert stroke; cognitive decline; delirium; clinical stroke; CABG surgery; near infrared spectroscopy; cerebral oxygenation
MeSH Terms: conditions — Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conducted a prospective observational pilot study to explore the incidence of peri-operative covert strokes (detected by brain MRI) and the potential impact on delirium and cognitive decline in post-operative cardiac surgery patients at the Hamilton General Hospital. This pilot study assessed the feasibility of a larger prospective international cohort study exploring this objective.

DETAILED DESCRIPTION:
Delirium and cognitive decline are common following cardiac surgery and increase the burden on patients and health care resources. Covert (sub-clinical) strokes are associated with these complications. The investigators conducted a prospective cohort pilot study enrolling consecutive cardiac surgery patients to receive a post-operative brain MRI and a series of questionnaires to assess for changes in cognition, physical function and delirium. Regional cerebral oxygen saturation (rSO2) was recorded during surgery with the use of near-infrared spectroscopy (NIRS) sensors placed on the patients' forehead. The primary aim was to determine the feasibility of conducting a larger study to establish an association between covert stroke and long-term cognitive decline in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 21 years old
2. Provide written informed consent
3. Scheduled to undergo isolated CABG through a median sternotomy approach
4. Have at least one of the following risk factors:

   1. Peripheral vascular disease (previous peripheral arterial bypass, amputation due to ischemia, ABPI <0.9, or previous AAA repair)
   2. Cerebrovascular disease (history of stroke, TIA, or carotid stenosis >70%)
   3. Renal insufficiency (eGFR <60 mL/min/1.73m2)
   4. Diabetes mellitus (on oral hypoglycemic agent(s) and/or insulin replacement)
   5. Urgent CABG (in-patient awaiting revascularization for ACS or MI)
   6. Recent smoker (within the last year)
   7. Left ventricular ejection fraction <35%

Exclusion Criteria:

1. Concomitant cardiac procedure with CABG Prior enrolment in this study
2. Emergency CABG surgery (immediate revascularization for hemodynamic instability)
3. Redo CABG
4. Circulatory arrest planned during the cardiac operation
5. Diagnosed dementia of any types
6. Contra-indication for DW MRI e.g. claustrophobia, unable to lie flat for the duration of the study, pacemaker or ICD in-situ, or other metal implants

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 21 years or more scheduled to undergo isolated coronary artery bypass grafting (CABG) surgery with a median sternotomy and at least one vascular risk factor.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 30 days
  Average recruitment rate per week
MRI completion | 30 days
  Total number of patients completing the brain MRI study
Lost to follow-up | 3 months
  Proportion of patients lost to follow-up at the end of the study

SECONDARY OUTCOMES:
Covert stroke | 30 days
  The proportion of patients experiencing covert stroke within 30 days of surgery
Clinical stroke | 30 days
  The proportion of patients experiencing clinical stroke 30 days after surgery
Cognitive decline (MoCA) | 30 days
  The proportion of patients experiencing cognitive decline 30 days after surgery using the Montreal Cognitive Assessment (MoCA).
Cognitive decline (DSST) | 30 days
  The proportion of patients experiencing cognitive decline 30 days after surgery using the Digit Symbol Substitution Test (DSST).
Physical function | 3 months
  The proportion of patients experiencing cognitive decline 30 days after surgery using the Standard Assessment of Global-activities in the Elderly (SAGE).
Delirium | day 2 to 30 day, whichever comes first
  The proportion of patients experiencing delirium between postoperative day 2 and discharge or 30 days, whichever comes first using the Confusion Assessment Method (CAM).

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mrkobrada M, Hill MD, Chan MT, Sigamani A, Cowan D, Kurz A, Sessler DI, Jacka M, Graham M, Dasgupta M, Dunlop V, Emery DJ, Gulka I, Guyatt G, Heels-Ansdell D, Murkin J, Pettit S, Sahlas DJ, Sharma M, Sharma M, Srinathan S, St John P, Tsai S, Gelb AW, O'Donnell M, Siu D, Chiu PW, Sharath V, George A, Devereaux PJ. Covert stroke after non-cardiac surgery: a prospective cohort study. Br J Anaesth. 2016 Aug;117(2):191-7. doi: 10.1093/bja/aew179. PMID 27440630
- [Background] NeuroVISION Investigators. Perioperative covert stroke in patients undergoing non-cardiac surgery (NeuroVISION): a prospective cohort study. Lancet. 2019 Sep 21;394(10203):1022-1029. doi: 10.1016/S0140-6736(19)31795-7. Epub 2019 Aug 15. PMID 31422895
- [Background] Indja B, Woldendorp K, Vallely MP, Grieve SM. Silent Brain Infarcts Following Cardiac Procedures: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2019 May 7;8(9):e010920. doi: 10.1161/JAHA.118.010920. PMID 31017035
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Vermeer SE, Longstreth WT Jr, Koudstaal PJ. Silent brain infarcts: a systematic review. Lancet Neurol. 2007 Jul;6(7):611-9. doi: 10.1016/S1474-4422(07)70170-9. PMID 17582361
- [Background] Smith EE, Saposnik G, Biessels GJ, Doubal FN, Fornage M, Gorelick PB, Greenberg SM, Higashida RT, Kasner SE, Seshadri S; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Functional Genomics and Translational Biology; and Council on Hypertension. Prevention of Stroke in Patients With Silent Cerebrovascular Disease: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Feb;48(2):e44-e71. doi: 10.1161/STR.0000000000000116. Epub 2016 Dec 15. PMID 27980126
- [Derived] Spence J, Lamy A, Bosch J, Thabane L, Gagnon S, Power P, Browne A, Murkin J, Devereaux PJ. Feasibility of studying the association between intraoperative regional cerebral oxygen saturation and postoperative functional decline (ReFUNCTION): a pilot sub-study of NeuroVISION-Cardiac Surgery. Can J Anaesth. 2020 Nov;67(11):1497-1506. doi: 10.1007/s12630-020-01777-3. Epub 2020 Aug 6. PMID 32767054